CLINICAL TRIAL: NCT03882801
Title: A Randomized Double Blind Clinical Trial to Evaluate the Effects of MK-7264 in Participants With Obstructive Sleep Apnea
Brief Title: Safety and Tolerability of Gefapixant (MK-7264) in Participants With Obstructive Sleep Apnea (MK-7264-039)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 7264-039; 2018-004099-37 (Other: EudraCT Number); MK-7264-039 (Other: MSD Protocol Number)
Record Dates: First submitted 2019-03-19; First posted 2019-03-20 (Actual); Results first posted 2020-11-19 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Gefapixant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1: Placebo -> Gefapixant (Experimental): In Period 1, participants receive a single oral dose of placebo matching gefapixant (MK-7264) every night at bedtime (QHS), for 7 days. In Period 2, participants receive a single oral dose of gefapixant (MK-7264) QHS, for 7 days. The two 7-day dosing periods are separated by a 7-day washout period.
  Interventions: Drug: Gefapixant; Drug: Placebo
- Sequence 2: Gefapixant -> Placebo (Experimental): In Period 1, participants receive a single oral dose of gefapixant (MK-7264) QHS for 7 days. In Period 2, participants receive a single oral dose of placebo matching gefapixant (MK-7264) QHS, for 7 days. The two 7-day dosing periods are separated by a 7-day washout period.
  Interventions: Drug: Gefapixant; Drug: Placebo

INTERVENTIONS:
Drug: Gefapixant — In Periods 1 and 2 (7 days each) participants receive 4 tablets (180 mg) of gefapixant (MK-7264) QHS.
  Other Names: MK-7264
Drug: Placebo — In Periods 1 and 2 (7 days each) participants receive 4 tablets of placebo QHS.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of multiple dose administration of gefapixant (MK-7264) in participants with moderate to severe obstructive sleep apnea (OSA). The primary hypothesis is that multiple dose administration of gefapixant (MK-7264) in participants with moderate to severe OSA reduces the Apnea Hypopnea Index (AHI) relative to placebo.

ELIGIBILITY:
Inclusion Criteria:

* International Classification of Sleep Disorders (ICSD-3) diagnosis of OSA, based on investigator's assessment of the obstructive sleep apnea (OSA) history and diagnostic interview which must include: Documented sleep study in the past that confirmed the OSA diagnosis without significant prior medical intervention.
* Apnea-Hypopnea Index (AHI) ≥ 20 events/hour at screening.
* No use of a positive airway pressure (PAP) device within the preceding 1 month or a dental appliance within the preceding 7 days prior to screening and is not allowed to use PAP or a dental appliance throughout the study (including washout intervals between treatment periods) and until the post-study visit.
* A baseline oxygen saturation via pulse oximetry (SpO2) ≥ 94% at screening to ensure that carotid body response to hyperoxia is not impaired.
* A body mass index (BMI) ≤ 35 kg/m^2 at the pre-study (Screening 1) visit.
* Judged to be in good health based on medical history, physical examination, vital sign measurements, and laboratory safety tests.
* No clinically significant abnormality on electrocardiogram (ECG)
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and is not a woman of childbearing potential (WOCBP) OR is a WOCBP and using an acceptable contraceptive method.
* A WOCBP must have a negative highly sensitive pregnancy test (urine as required by local regulations) within 72 hours before the first dose of study intervention.
* If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required.
* The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* A consistent sleep-wake schedule that is not subject to any other unusual changes in sleeping routine (i.e., bedtimes and wake times do not vary more than 1-2 hours except on rare occasions).
* Able to maintain sleep for at least 4 consecutive hours based on self-report.

Exclusion Criteria:

* Other than OSA, has evidence of another clinically significant, active pulmonary disorder such as bronchiectasis, emphysema, or asthma documented by history, physical examination, or chest x-ray.
* A history within the past 6 months prior to the pre-study visit or current evidence of an unstable or clinically significant cardiovascular disorder, including but not limited to: acute coronary syndrome, unstable angina, congestive heart failure, cardiogenic syncope, cardiomyopathy, any symptomatic arrhythmia, orthostatic hypotension, uncontrolled hypertension, chronic kidney disease, kidney transplant
* Abnormal pre-randomization laboratory values for alanine transaminase > 1.5 x the upper limit of normal (x ULN), aspartate transaminase > 1.5 x ULN, direct bilirubin > 1.5 x ULN, serum creatinine of > 2 mg/dL
* A history or diagnosis of any of the following conditions, in the opinion of the investigator: narcolepsy (with or without cataplexy) or Idiopathic hypersomnia, circadian rhythm sleep disorder, parasomnia including nightmare disorder, sleep terror disorder, sleepwalking disorder, and rapid eye movement (REM) behavior disorder, periodic limb movement (PLM) disorder, restless legs syndrome, chronic insomnia
* A WOCBP who has a positive urine or serum pregnancy test within 24 hours before the baseline 1 of study intervention.
* A history of clinically significant or poorly-controlled endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* Mentally or legally incapacitated, or has significant emotional problems at the time of pre-study screening
* A history or current evidence of any condition, therapy, lab or ECG abnormality or other circumstances that might confound the results of the study, or interfere with the participant's participation for the full duration of the study.
* Any history of a neurological disorder, including but not limited to seizure disorder (other than single episodes of childhood febrile seizures), stroke, transient ischemic attack, multiple sclerosis, cognitive impairment, or significant head trauma with sustained loss of consciousness within the last 10 years.
* A history of significant multiple and/or severe allergies (e.g., food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (i.e., systemic allergic reaction) to prescription or non-prescription drugs or food.
* A history of anaphylaxis or cutaneous adverse drug reaction (with or without systemic symptoms) to sulfonamide antibiotics or other sulfonamide-containing drugs.
* Positive for hepatitis B surface antigen, hepatitis C antibodies or HIV.
* A history of cancer (malignancy) with some exceptions including adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix or; and other malignancies that have been successfully treated with appropriate follow up and therefore unlikely to recur for the duration of the study, in the opinion of the investigator and with agreement of the Sponsor (e.g., malignancies that have been successfully treated ≥ 10 years prior to the pre-study [screening] visit).
* An estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m^2 based on the Cockcroft-Gault (CG) Equation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- United States (4):
  - MD Clinical ( Site 0004), Hallandale, Florida
  - Research Centers of America, LLC ( Site 0002), Hollywood, Florida
  - Neurotrials Research, Inc. ( Site 0001), Atlanta, Georgia
  - Clinilabs, Inc. ( Site 0005), New York, New York
- Universitair Ziekenhuis Gent ( Site 0012), Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Robbins JA, Sands S, Maganti L, Crumley T, Fox-Bosetti S, Hussain A, Schwartz H, Safirstein B, Ahmad M, Dragone L, Nussbaum J, Kushida C, Iwamoto M, Stoch SA. Gefapixant as a P2X3 receptor antagonist treatment for obstructive sleep apnea: a randomized controlled trial. J Clin Sleep Med. 2024 Dec 1;20(12):1905-1913. doi: 10.5664/jcsm.11272. PMID 39069967

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 3 centers in a single country
Pre-assignment Details: 24 participants were randomized and enrolled, 23 were administered with at least one dose of study drug, 1 participant was never dosed.
Groups:
- Placebo Then Gefapixant 180 mg: Placebo once daily at bedtime (QHS) oral for 7 days in Period 1 followed by a 7-day washout period and then Gefapixant, 180 mg, QHS, oral for 7 days in Period 2.
- Gefapixant 180 mg Then Placebo: Gefapixant, 180 mg, QHS, oral for 7 days in Period 1 followed by a 7-day washout period and then placebo, QHS, oral for 7 days in Period 2.
Period: Period 1
Arm/Group | Placebo Then Gefapixant 180 mg | Gefapixant 180 mg Then Placebo
Started | 12 | 12
Treated | 11 (1 participant did not receive any dose of study drug) | 12
Completed | 10 | 10
Not Completed | 2 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Non-compliance with study drug | 1 | 1
Not completed — Never treated with study drug | 1 | 0
Period: Washout Period
Arm/Group | Placebo Then Gefapixant 180 mg | Gefapixant 180 mg Then Placebo
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Period 2
Arm/Group | Placebo Then Gefapixant 180 mg | Gefapixant 180 mg Then Placebo
Started | 10 | 9
Completed | 10 | 8
Not Completed | 0 | 1
Not completed — Non-compliance with study drug | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Gefapixant 180 mg | Gefapixant 180 mg Then Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.7 (7.0) | 56.4 (7.9) | 55.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Apnea-Hypopnea Index (AHI) Change From Baseline as Calculated From Polysonagraphy (PSG)
Description: The apnea-hypopnea index (AHI) is the sum of the apnea and hypopnea indices for each participant. The apnea index for each participant is calculated as the number of apneas divided by the total sleep time. The hypopnea index for each participant is calculated as the number of hypopneas divided by the total sleep time. These measurements are collected from polysonagraphs (PSGs), which are diagnostic sleep studies that collect electroencephalogram (EEG), electrooculograph (EOG), electromyogram (EMG), electrocardiogram (ECG), airflow, respiratory effort, oximetry, and sleep position data. Baseline AHI measurements in each period are obtained on Day -1. Individual AHI fold-change from baseline in each treatment period are calculated as the ratio of on-treatment AHI to baseline AHI.
Time Frame: Day-1 at Baseline and Day 7 of each treatment period
Population: Analysis population consisted of all randomized participants who received at least 1 dose of study drug, were compliant with the study procedure and had available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Groups:
- Placebo: Placebo once daily at bedtime (QHS) taken orally for 7 days
- Gefapixant 180 mg: Gefapixant, 180 mg, QHS, taken orally for 7 days
Arm/Group | Placebo | Gefapixant 180 mg
Number analyzed (Participants) | 18 | 19
ratio | 0.86 [0.68 to 1.09] | 0.97 [0.74 to 1.27]
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 180 mg; Test type: Superiority; Least Square Geometric Means Ratio = 0.92, 90% CI 2-sided [0.73 to 1.17] — Back transformed least squares mean and confidence interval from linear mixed effects model performed on natural log-transformed values

2. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE) During the Study
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the product, is also an AE.
Time Frame: Up to 14 days after last dose of study drug (Up to 35 days)
Population: Any participant who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Gefapixant 180 mg
Number analyzed (Participants) | 20 | 22
Participants | 2 | 13

3. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 2
Time Frame: Up to 21 days
Population: Any participant who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Gefapixant 180 mg
Number analyzed (Participants) | 20 | 22
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 14 days after last dose of study drug (Up to 35 days)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated, and/or related with the study drug. Any worsening of a preexisting condition which is temporally associated with the study drug, is also an AE. All-Cause Mortality table includes all randomized participants. Serious Adverse Events and Other Adverse Events tables include all randomized participants who received ≥1 dose of study drug.
Groups:
- Screening: Screening
- Gefapixant: Gefapixant 180 mg QHS taken orally for 7 days
- Post Trial: Post trial
Arm/Group | Screening | Gefapixant | Placebo | Post Trial
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/22 | 0/20 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22 | 0/20 | 0/24
Other Adverse Events (participants affected / at risk) | 2/24 | 13/22 | 2/20 | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screening (N=24) | Gefapixant (N=22) | Placebo (N=20) | Post Trial (N=24)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysphoria (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Physical assault (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with standard editorial and ethical practice, the Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/01/NCT03882801/Prot_SAP_000.pdf